## A single center randomized prospective study on the criteria for lymph node sorting for pathological examination after curative surgery for gastric cancer

(DJY001 Trail)

**Edition Number: 1.0** 

**Edition Generation Date: Qct 30, 2017** 

Principal Investigator: Jingyu Deng and Han Liang

Research Institute: Cancer Hospital & Institute of Tianjin Medical University

## Statistical Analysis Plan

Continuous variables are expressed as mean and range. Clinicopathological characteristics significantly related to patients' survival were evaluated with reference to statistics obtained by the Kaplan-Meier method for calculating the OS, and Cox proportional hazards analysis was performed for the multivariate survival analysis. The Bayesian information criterion (BIC) value within a Cox proportional hazard regression model were calculated for each category to measure its discriminatory ability. The case-control matched logistic regression (using the forward stepwise procedure, and the ratio between the number of cases and the number of controls=1:1) was used to directly compare the prognostic prediction superiority of the fine sorting lymph node method to that of the regional sorting lymph node method in various subgroups of patients. Significance was defined as a P value < 0.05. All statistical analyses were performed using PASW 18.0 software.